CLINICAL TRIAL: NCT01013688
Title: Efficiency of Radiofrequency Ablation for Surgical Treatment of Chronic Atrial Fibrillation With Rheumatic Valve Disease
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: China National Center for Cardiovascular Diseases, China National Center for Cardiovascular Diseases
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Wangxin
Record Dates: First submitted 2009-11-11; First posted 2009-11-16 (Estimated); Last update posted 2009-11-18 (Estimated); Status verified 2009-11

CONDITIONS: Rheumatic Valve Disease; Atrial Fibrillation
Keywords: Radiofrequency ablation; Maze; Atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- left atrial RF ablation groups (Experimental): Excised the left atrial appendage Encircling the left pulmonary veins and an extension to the posterior mitral valve annulus From the left atrial appendage to the left superior pulmonary vein A connecting line between both islands of pulmonary veins From the middle of the mitral valve ablation line down towards the base of the atria ligament of Marshall
  Interventions: Procedure: Cardioblate® Surgical Ablation System
- Bi-atrial radiofrequency ablation group (Experimental): In the basis of left atrial group,excised the right atrial appendage; from the amputated right atrial appendage towards the inferior vena cava; from the midterm of interatrial septum to the AV groove; ablation between the superior and inferior caval cannulation sites; radiofrequency ablation for Waterston's groove
  Interventions: Procedure: Cardioblate® Surgical Ablation System
- Amiodarone group (No Intervention): No radiofrequency ablation procedure during the valve surgery; Amiodarone 200 mg/day for 12 months after surgery

INTERVENTIONS:
Procedure: Cardioblate® Surgical Ablation System — Using Cardioblate® Surgical Ablation System to perform left atrial or bi-atrial radiofrequency ablation procedure during valve surgery
  Other Names: radiofrequency
  Arms: Bi-atrial radiofrequency ablation group; left atrial RF ablation groups

SUMMARY:
The purpose of this study is to determine whether concomitant radiofrequency Maze procedure for surgical treatment of chronic atrial fibrillation with rheumatic valve disease could provide better sinus rhythm control, improved cardiac hemodynamic status and decreased thromboembolism events and to compare if biatrial is better than left atrial procedure? 150 rheumatic valve patients with chronic atrial fibrillation (AF) having concomitant valve surgery were randomized to three groups: left atrial ablation group, bi-atrial ablation group, and Amiodarone group. All patients were scheduled followed up before discharge and at 3rd, 6th and 12th postoperative months. Standard 12-lead electrocardiography (ECG), 24-hour Holter and transthoracic echocardiography were used to determine the rhythm and cardiac hemodynamic status.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether concomitant radiofrequency Maze procedure for surgical treatment of chronic atrial fibrillation with rheumatic valve disease could provide better sinus rhythm control,improved cardiac hemodynamic status and decreased thromboembolism events and to compare if biatrial is better than left atrial procedure?

150 patients with chronic AF having concomitant cardiac surgery will be enrolled. Patients will underwent bi-atrial radiofrequency,left atrial radiofrequency or no radiofrequency procedure randomly. All the patients will receipt amiodarone 200 mg/day for 12 months postoperatively.

All patients were scheduled followed before discharge and at 3rd, 6th and 12th postoperative months.The following diagnostic procedures were performed

1. Standard 12-lead electrocardiography
2. Holter-ECG
3. Transthoracic echocardiography

ELIGIBILITY:
Inclusion Criteria:

1. Patients with atrial fibrillation secondary to definite rheumatic valve disease
2. At least six months and no longer than 5 years of chronic atrial fibrillation
3. Age >=18 years and <=70 Patients who can give informed consent themselves in writing
4. No contraindication for amiodarone
5. Negative pregnancy test (in women with childbearing potential)

Exclusion Criteria:

Any one of the following exclusion criteria is sufficient to disqualify a patient from the study

1. Left atrial diameter(LAD)>=70mm
2. Left ventricular eject fraction(LVEF)<=30%
3. Atrial thrombus
4. Contraindication for anticoagulation therapy
5. Less than 6 months since last episode of cerebral infarction
6. Emergency operation
7. Patients with a malignant tumor
8. Pregnant or nursing patients, those who may be pregnant, or those who plan on becoming pregnant before the end of the study period.
9. Any other reason that the Clinical Supervisors or Clinical Researchers may have for considering a case unsuitable for the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2008-03; Primary Completion 2009-05 (Estimated); Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
At 3rd, 6th and 12th month's follow-up, to evaluate the rhythm status by ECG and 24-hour Holter and cardiac hemodynamic status by transthoracic echocardiography | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Shengshou Hu, Study Director — National center for cardiovascular disease ,china
Locations (1):
- Fuwai cardiovascular disease hospital, Beijing, China

REFERENCES:
- [Derived] Wang X, Wang X, Song Y, Hu S, Wang W. Efficiency of radiofrequency ablation for surgical treatment of chronic atrial fibrillation in rheumatic valvular disease. Int J Cardiol. 2014 Jul 1;174(3):497-502. doi: 10.1016/j.ijcard.2014.03.153. Epub 2014 Mar 29. PMID 24820759